CLINICAL TRIAL: NCT04298892
Title: Integrated Multiomics and Multilevel Characterization of Haematological Disorders and Malignancies
Acronym: INTHEMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Azienda Unità Sanitaria Locale della Romagna (Other)
Responsible Party: Sponsor
Other Study IDs: IRSTB100
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-09

CONDITIONS: Haematologic Disease; Haematological Malignancy
Keywords: Hematologic malignancies; omics; integrated; translational
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Fresh peripheral blood, bone marrow, urine, bone biopsy, lymph node biopsy, cerebrospinal, ascites, pericardial and pleural fluid. All samples will be collected according to clinical practice. In addition, a saliva sample will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hematologic disorder or malignancy
  Interventions: Other: clinical data and sample collection

INTERVENTIONS:
Other: clinical data and sample collection — Patients with hematologic malignancies and disorders will be asked to donate part of the samples collected as per clinical practice for the management of their disease for the aims of this study. In addition, patients will be asked to donate one oral swab sample, and urine samples. Collection of these additional samples is a non-invasive procedure with no associated risks for patients. Clinical data (demographics including ethnicity, stage of disease, concise treatment history, cytogenetic reports, and molecular data if available, as routinely performed during diagnosis procedures) will be collected.

SUMMARY:
Exploratory multicenter, non-interventional, translational, retrospective and prospective study. All patients with a diagnosis of hematologic disorder or malignancy for whom biological samples and clinical data are available may be included in this study, after obtaining informed consent

DETAILED DESCRIPTION:
Hematological malignancies account for approximately 9.5% of newly diagnosed cancers every year and their incidence shows an exponential rise after the age of 40. Since life expectancy is dramatically and continuously increasing worldwide, hematological diseases promise to become a substantial burden for the health care systems of the European society. The management of hematological malignancies is further complicated by the high level of disease heterogeneity in terms of pathogenic and molecular mechanisms. Due to the high level of heterogeneity in terms of cytogenetic, genetic, epigenetic, transcriptional, post-transcriptional and metabolic alterations, an accurate molecular classification of hematological diseases is needed to improve clinical outcomes and patients' management. This is an exploratory multicenter, non-interventional, translational, retrospective and prospective study. All patients with a diagnosis of hematologic disorder or malignancy for whom biological samples and clinical data are available may be included in this study, after obtaining informed consent. The primary objective is to improve our knowledge of the pathogenic mechanisms driving malignant disorders and transformation. The secondary objectives aim to improve diagnosis and stratification of onco-hematological patients and study drug response at preclinical level. After signing informed consent to the study, each patient will donate part of the samples (peripheral blood, bone marrow, biopsies) collected as per routine clinical practice for the management of their disease.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study
2. Male or Female, aged >18 years
3. Patients with histologically confirmed diagnosis of one of the following haematological diseases: monoclonal gammopathy of undetermined significance (MGUS), idiopathic cytopenia of undetermined significance (ICUS), clonal cytopenia of undetermined significance (CCUS), clonal hematopoiesis of indeterminate potential (CHIP) or hematological malignancies: Peripheral T-cell Lymphomas (PTCL), B- and T-Lymphoblastic Leukemias / Lymphomas (ALL), Burkitt Lymphoma (BL), B and T cell lymphoma, Acute Myeloid Leukemia (AML), Myeloproliferative Disease (Polycythemia Vera (PV), Essential Thrombocythemia (ET), Monocytic Leukemia), Chronic Lymphocytic Leukemia (CLL), Chronic Myeloid Leukemia (CML), Myelofibrosis, Myelodysplasia (MDS) including Macrocytic Anemia, Sideroblastic Anemia and Non-Neoplastic Hematologic Disease, Systemic Mastocytosis, Multiple Myeloma (MM), Plasma Cell Disease.
4. Available clinical data (demographics including ethnicity, stage of disease, concise treatment history, cytogenetic reports, and molecular data if available, as routinely performed during diagnosis procedures);
5. For the retrospective part of the study: availability of biological samples collected for routine diagnostics/therapeutic procedures and stored as appropriate, per laboratory standard procedures.

Exclusion Criteria:

* Patients included in clinical trials may be enrolled in this explorative study, except where otherwise clearly indicated in the experimental protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with haematological malignancy or disorder (see inclusion criteria) treated in the participating centers will be considered for enrollment. Patients can be enrolled at diagnosis or at relapse. Samples will be collected before treatment, during treatment whenever possible, at follow-up, at remission and at each relapse.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
haematologic diseases characterization | up to 5 years
  To improve our knowledge of the pathogenic mechanisms driving malignant disorders and transformation in different subgroups, defined by molecular, metabolic, proteomic, imaging, preclinical and clinical data integration

SECONDARY OUTCOMES:
Ex vivo Response/resistance | up to 5 years
  To define response/resistance to ex vivo drug treatments;
toxicity biomarkers identification | up to 5 years
  To identify biomarkers of drug-related toxicity;
Biological and molecular features | up to 5 years
  To investigate association between biological and molecular features with patient's clinical features.
Minimal residual disease (MRD) | up to 5 years
  To investigate recurrence/minimal residual disease patterns after treatments
Prognostic and early diagnostic biomarkers | up to 5 years
  To identify novel biomarkers for early diagnosis (e.g. predictive of transformation from a pre-malignant to an overt malignant phase) and prognosis.
identification of circulating and tissue molecular markers. | up to 5 years
  To improve the diagnostic work-up of haematological disease, thus enlarging the fraction of patients suitable for curative treatments through the identification of circulating and tissue molecular markers.
technological advancement | up to 5 years
  To provide a technological advancement potentially applicable to the national health system, when properly validated in appropriate patients' subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Prof, Study Director — IRST IRCCS; Alessandro Lucchesi, MD, Principal Investigator — IRST IRCCS
Locations (26):
- Italy (26):
  - Irst Irccs, Meldola, FC
  - C.R.O.B. - I.R.C.C.S., Rionero in Vulture, Potenza
  - AOU Città della Salute e della scienza di Torino, Torino, TO
  - Centro di Riferimento Oncologico - CRO Irccs, Aviano
  - A.O.U. Consorziale policlinico Giovanni XXIII di Bari, Bari
  - IRCSS Istituto Tumori, Bari
  - Ospedale A. Perrino, Brindisi
  - Ospedale Santa Croce e Carle, Cuneo
  - IRCCS Osp. Policlinico San Martino, Genova
  - Istituto Giannina Gaslini, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - IEO, Milan
  - Istituto Nazionale Tumori Di Napoli Irccs, Napoli
  - AORN " A. Cardarelli", Napoli
  - AUO San Luigi Gonzaga, Orbassano
  - Irccs Iov, Padua
  - AOU "P. Giaccone", Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - P.O. Santo Spirito, Pescara
  - UO Hematology, Ospedale S. Maria delle Croci, Ravenna
  - Arcispedale S. Maria Nuova - AUSL IRCCS, Reggio Emilia
  - UO Hematology Ospedale Infermi, Rimini
  - IRCCS Fondazione Policlinico Universitario A. Gemelli, Roma
  - AOU" San Giovanni di Dio e Ruggi d'Aragona", Salerno
  - AO Ordine Mauriziano, Torino
  - Ospedale Ca' Foncello Treviso, Treviso

IPD SHARING:
Plan to Share IPD: No